CLINICAL TRIAL: NCT00037609
Title: Phase I-II Study to Evaluate Safety, Efficacy and Pharmacokinetic Interactions Between Capecitabine (XELODA) and Exisulind (APTOSYN) in Patients With Metastatic Breast Cancer
Brief Title: Safety, Efficacy and Pharmacokinetic Between Capecitabine and Exisulind in Metastatic Breast Cancer Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Cell Pathways (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID00-049
Record Dates: First submitted 2002-05-17; First posted 2002-05-20 (Estimated); Last update posted 2012-10-24 (Estimated); Status verified 2012-10

CONDITIONS: Breast Neoplasms; Metastases, Neoplasm
Keywords: Metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Capecitabine; sulindac sulfone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Capecitabine + Exisulind (Experimental): Capecitabine 1000 mg/m^2 taken by mouth twice daily. Exisulind 125 mg taken by mouth twice daily.
  Interventions: Drug: Capecitabine; Drug: Exisulind

INTERVENTIONS:
Drug: Capecitabine — 1000 mg/m^2 taken by mouth twice daily.
  Other Names: Xeloda
Drug: Exisulind — 125 mg taken by mouth twice daily.
  Other Names: Aptosyn

SUMMARY:
The primary objective of the phase I study is to determine a safe dose for combination therapy with capecitabine and exisulind. A secondary objective is to assess pharmacokinetic interactions between the two drugs and assess the biological activity of exisulind.

The primary objective of the Phase II part of this study is to assess the anti-tumor activity of this combination therapy measured by objective tumor response. Secondary end points also assessed will be toxicity of therapy, duration of response and time to progression.

DETAILED DESCRIPTION:
Rationale for this study:

Capecitabine is approved by the Food and Drug Administration (FDA) as 2nd or 3rd line chemotherapy for patients with metastatic breast cancer who previously have failed both anthracycline and taxane chemotherapy. Capecitabine produces objective tumor response of around 20% with a median duration of response of 32 weeks in these patients (1). These results indicate that improvements in the treatment of anthracycline and taxane resistant breast cancer are needed. Exisulind (sulindac sulfone, FGN-1, APTOSYNTM) is a sulfone metabolite of sulindac, a widely used nonsteroidal anti-inflammatory (NSAID) drug. Sulindac sulfone lacks inhibitory activity on the two isoforms of cyclooxygenase, COX 1 and COX 2, and is devoid of gastrointestinal and renal toxicity that is associated with NSAIDs. Exisulind selectively stimulates programmed cell death in a variety of neoplastic cells including colon, prostate, and mammary epithelial cells without affecting normal cells (2,3). Exisulind inhibits the growth of breast cancer cell lines in vitro and also inhibits chemically-induced mammary carcinogenesis in rats (4,5). The drug is also synergistic with a diverse group of cytotoxic compounds including cisplatin, taxanes and retinoids (6). Exisulind exerts its effects by inhibiting a novel phosphodiesterase that belongs to the PDE5 family which specifically degrades cGMP (7). Inhibition of this enzyme results in a rise in intracellular cGMP levels and leads to apoptosis through yet unknown mechanism. Exisulind also inhibits transcription factor NF-kB (8). The NF-kB pathway is activated by cellular stress including exposure to inflammatory cytokines, cytotoxic agents and oxidative stress (9). It is believed that activation of NF-kB protects from cell death, therefore, inhibition of this transcription factor may contribute to the proapoptotic, chemotherapy potentiating effect of exisulind.

Exisulind selectively promotes apoptosis in neoplastic cells whereas chemotherapeutic drugs induce programmed cell death in a non-selective manner. We hypothesize that combination of the 2 drugs will increase response rates by selectively augmenting the cytotoxic activity of chemotherapy. Furthermore, continuous maintenance treatment, between chemotherapy doses, with a minimally toxic drug that selectively induces apoptosis of cancer cells may improve response duration and ultimately may translate into improved survival and better quality of life. Each drug alone has an established maximum tolerated dose in humans. However, the combination of exisulind and capecitabine has not been tested. This phase I-II study is proposed to test safety and efficacy of this combination in patients with metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria

Each patient must meet all these criteria in order to be considered for enrollment in the Phase I study:

* Histologically confirmed breast cancer and either clinical, radiological or laboratory evidence of metastatic disease.
* Patients must have received both anthracycline-containing and taxane chemotherapy either as adjuvant treatment or therapy for metastatic breast cancer.
* There is no limit on prior chemotherapy regimens or hormonal therapies received.
* Concomitant bisphosphonate treatment is allowed for patients with bone metastases.
* Patients must have recovered from acute toxic effects of any prior therapy including surgery and radiation.
* Zubrod performance status < 2. (See Appendix A)
* Adequate bone marrow function: platelets > 100,000/mm3, ANC > 1500 cells/mm3, hemoglobin > 8g/dl.
* Normal renal function: creatinine < 2.0 mg/dl.
* Adequate liver function: Bilirubin < 1.5 mg/dL. Transaminases (SGOT) or LDH, and alkaline phosphatase must be <1.5 x of the upper limit of normal in the absence of bone or liver metastasis, or <2.5 x of the upper limit of normal in the presence of radiologically apparent liver metastasis or bone metastasis, respectively.
* Female patients must be of non-childbearing potential or non-lactating and using adequate contraception. Beta-HCG will be checked in premenopausal patients if clinically indicated.
* Patients with brain metastases whose disease remained stable for more than 6 months after completing therapy to the brain are eligible.
* Written informed consent.

In addition to the above, patients participating in the Phase II portion of this study:

Must have bidimensionally measurable or evaluable disease. Lytic lesions seen on plain radiographs will be considered evaluable in conjunction with bone scan abnormalities. Bone scan abnormalities alone, pure blastic bone metastases or irradiated lesions are not considered measurable or evaluable and will not be accepted. Also, pleural or peritoneal effusions will not be considered evaluable disease.

Exclusion Criteria

A patient must not be enrolled if any of the following criteria applies:

* Known hypersensitivity to sulindac (CLINORIL).
* Known hypersensitivity or contraindications to capecitabine (XELODAR) including prior therapy with capecitabine.
* Clinical or laboratory evidence of significant liver disease.
* Concomitant treatment with cytotoxic agents other than capecitabine or participation in any other investigational study.
* Uncontrolled psychiatric, or social (addictive) disorders that would preclude obtaining informed consent or patient participation in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2001-01; Primary Completion 2003-02 (Actual); Study Completion 2003-02 (Actual)

PRIMARY OUTCOMES:
Response Rate | Blood tests done every week for first 6 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Lajos Pusztai, MD, DPHIL, Study Chair — UT MD Anderson Cancer Center
Locations (1):
- University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org